CLINICAL TRIAL: NCT05211583
Title: Evaluation of Serum Hormone Levels Referenced to Ovulation in Subfertile Women With Regular Menses
Brief Title: Serial Progesterone Level Measurements During the Menstrual Cycle in Subfertile Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turgut Aydın (Other)
Responsible Party: Sponsor-Investigator, Turgut Aydın, Associate Clinical Professor, Acibadem University
Organization: Acibadem University (Other)
Other Study IDs: Progesterone
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Subfertility, Female; Ovulation Disorder
Keywords: ovulation; progesterone; ovulatory dysfunction; subfertility
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- subfertile women: Subfertile women with regular menses (menstrual cycle length range from 21 to 35 days) will be examined by transvaginal ultrasonography at menstruation, before the anticipated date of ovulation and after ovulation. Serum hormone levels will be measured at menstruation, before ovulation and after ovulation with a serial manner.
  Interventions: Diagnostic Test: Serum progesterone levels

INTERVENTIONS:
Diagnostic Test: Serum progesterone levels — In order to show change of serum progesterone levels, serial venous blood sampling will be done and also transvaginal ultrasonography will be performed to show ovulation.

SUMMARY:
Ovulatory dysfunction is identified in 15% of all infertile couples and it accounts for 40% of female infertility. Ovulatory dysfunction may be more subtle in women with regular menses. Detecting the day of ovulation is necessary for optimizing natural conception, diagnosis of cycle disturbances and also timing for embryo transfer in natural cycle frozen-thawed embryo transfers. In order to diagnose ovulatory dysfunction, ovulation physiology and change of reproductive hormones during the menstrual cycle should be understood. In the present study we aimed to evaluate serial serum hormonal cut-off levels referenced to ovulation in subfertile women with regular menses.

ELIGIBILITY:
Inclusion Criteria:

* women that have regular menses (menstrual cycle length 21-35 days)
* women who will come visits regularly
* women that are trying to conceive more than 1 year if women age is less than 35 years or more than 6 months if women age is >35 years

Exclusion Criteria:

* women who do not menstruate regularly
* women that use hormonal contraception
* women who take drugs that will interfere with steroid hormone metabolism

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will be selected from women who attended to Acıbadem University Atakent Hospital Infertility Clinic for evaluation of infertility.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change of serum progesterone levels referenced to ovulation | Progesterone levels will be measured serially when dominant follicule reaches 17 mm in diameter and after that 1-2 days interval until to ovulation; 1 week after ultrasound and hormone-detected ovulation
  Serum progesterone levels will be measured when dominant follicule is 17 mm in diameter and then serial measurements of hormones will be done and ovulation will be detected both hormonally and ultrasonographically. The range of serum progesterone will be reported referenced to ovulation.
Change of reproductive hormone levels referenced to ovulation | Estradiol and LH levels will be measured serially when dominant follicule reaches 17 mm in diameter and after that 1-2 days interval until to ovulation.
  Serum estradiol and luteinising hormone (LH) levels will be measured when dominant folicule is 17 mm in diameter and then serial measurements of hormones will be done and ovulation will be detected both hormonally and ultrasonographically. The ranges for serum hormones will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Aydın, Principal Investigator — Acibadem University
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No